CLINICAL TRIAL: NCT05021666
Title: A Phase 1, Double-blind, Randomized, Placebo-controlled, Single- and Multiple-dose Escalating Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of PB-718 Following Subcutaneous Administration in Healthy Subjects
Brief Title: A Phase 1, Double-blind, Randomized, Placebo-controlled, Single- and Multiple-dose Escalating Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PegBio Co., Ltd. (Other)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: PB718-001
Record Dates: First submitted 2021-08-16; First posted 2021-08-25 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Intervention Model Description: In Part A, 48 subjects will be studied in 6 groups (Groups A1 to A6), with each group consisting of 8 subjects.
  In Part B, 32 subjects will be studied in 4 groups (Groups B1 to B4), with each group consisting of 8 subjects Following review of the safety, tolerability, and PK data, additional dose groups may be added to the study. Up to 3 further groups of 8 subjects (6 PB-718: 2 placebo) may be included in each of Parts A and B.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The Investigator and other members of staff involved with the study will remain blinded to the treatment randomization code during the assembly procedure. The placebo solution will be identical in appearance to the PB-718.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Group A1 (Experimental): PB-718 vs placebo
  Interventions: Drug: Placebo; Drug: PB 718
- Group A2 (Experimental): PB-718 vs placebo
  Interventions: Drug: Placebo; Drug: PB 718
- Group A3 (Experimental): PB-718 vs placebo
  Interventions: Drug: Placebo; Drug: PB 718
- Group A4 (Experimental): PB-718 vs placebo
  Interventions: Drug: Placebo; Drug: PB 718
- Group A5 (Experimental): PB-718 vs placebo
  Interventions: Drug: Placebo; Drug: PB 718
- Group A6 (Experimental): PB-718 vs placebo
  Interventions: Drug: Placebo; Drug: PB 718
- Group B1 (Experimental): PB-718 vs placebo
  Interventions: Drug: Placebo; Drug: PB 718
- Group B2 (Experimental): PB-718 vs placebo
  Interventions: Drug: Placebo; Drug: PB 718
- Group B3 (Experimental): PB-718 vs placebo
  Interventions: Drug: Placebo; Drug: PB 718
- Group B4 (Experimental): PB-718 vs placebo
  Interventions: Drug: Placebo; Drug: PB 718

INTERVENTIONS:
Drug: Placebo — matching placebo
Drug: PB 718 — dose in the next group will be determined following a review of data from the previous group

SUMMARY:
This will be a randomized, double-blind, placebo-controlled, single- and multiple SC dose escalating study conducted in 2 parts.

DETAILED DESCRIPTION:
A Phase 1, double-blind, randomized, placebo-controlled, single and multiple-dose escalating study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of PB-718 following subcutaneous administration in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and willing to sign an ICF and to abide by the study restrictions.
2. Males or females, of any race, between 18 and 55 years of age, inclusive.
3. Male subjects will weigh at least 50 kg, and female subjects will weigh at least 45 kg. Body mass index between 20.0 and 30.0 kg/m2 (Part A) or 25.0 to 50.0 kg/m2 (Part B), inclusive.
4. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at Screening and Check-in/predose as assessed by the Investigator (or designee).

Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, renal, hematological, pulmonary, cardiovascular or other heart disease, gastrointestinal, urinary/prostatic, neurological, respiratory, endocrine, or psychiatric disorder, or glaucoma, as determined by the Investigator (or designee).
2. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
3. Liver disease or liver injury, as indicated by abnormal liver function tests (e.g. serum bilirubin, direct bilirubin, ALT, AST, γ-GT, or ALK exceeding the ULN) at Screening or Baseline which may be repeated for confirmation per the Investigators discretion at Screening and Check-in.
4. History of multiple endocrine neoplasia type 2 or an abnormal thyroid function test (thyroid stimulating hormone, triiodothyronine, thyroxine) at Screening or Baseline.
5. Fasting plasma glucose greater than ≥126 mg/dL at Baseline.
6. Hemoglobin A1c value >6.5%
7. History of chronic or acute pancreatitis, or amylase or lipase exceeding 2 × ULN at Screening or Baseline. -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From Group A1 until Group B4. The study duration for each subject in Part A will be approximately 8 weeks. The study duration for each subject in Part B will be approximately 11 weeks.
  Incidence, causality, and severity of AE. The condition of each subject will be monitored from the time of signing the ICF to Final Discharge from the study. Subjects will be observed for any signs or symptoms and asked about their condition by open questioning, such as "How have you been feeling since you were last asked?", at least once each day while resident at the study site and at each study visit. Subjects will also be encouraged to spontaneously report AEs occurring at any other time during the study.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile | From Group A1 until Group B4. The study duration for each subject in Part A will be approximately 8 weeks. The study duration for each subject in Part B will be approximately 11 weeks.
  AUC (area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration) from time zero to the time of the last quantifiable concentration (AUC0-tlast)
Pharmacokinetic (PK) profile | From Group A1 until Group B4.The study duration for each subject in Part A will be approximately 8 weeks. The study duration for each subject in Part B will be approximately 11 weeks.
  Cmax (maximum observed plasma concentration)
Pharmacokinetic (PK) profile | From Group A1 until Group B4. The study duration for each subject in Part A will be approximately 8 weeks. The study duration for each subject in Part B will be approximately 11 weeks.
  Tmax (time of the maximum observed plasma concentration)
Pharmacokinetic (PK) profile | From Group A1 until Group B4. The study duration for each subject in Part A will be approximately 8 weeks. The study duration for each subject in Part B will be approximately 11 weeks.
  terminal disposition phase rate constant (λz)

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Coleman, MD, Principal Investigator — Daytona Beach CRU
Locations (1):
- Covance Clinical Research Unit Inc., Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided